CLINICAL TRIAL: NCT06688773
Title: THE EFFECT OF PROGRESSIVE RELAXATION EXERCISES ON COMFORT AND ANXIETY LEVEL OF PATIENTS WITH LUMBAR DISC HERNIATION SURGERY: CLINICAL TRIAL
Brief Title: THE EFFECT OF RELAXATION EXERCİSE ON COMFORT AND ANXIETY IN HERNIATED LUMBAR DISC SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Didem Ayhan, Associate Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BOEU-RSPH-BC-01
Record Dates: First submitted 2024-11-07; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Disc Herniation
Keywords: Anxiety; comfort level; nursing; lumbar disc herniation; progressive relaxation exercises
MeSH Terms: conditions — Intervertebral Disc Displacement; Anxiety Disorders | interventions — Prostaglandins E

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- progressive relaxation exercises group (Experimental)
  Interventions: Behavioral: Progressive relaxation exercise
- Control group (Other): Implementation of standart postoperative care in the clinical setting.
  Interventions: Other: Control group: Standart nursing care group

INTERVENTIONS:
Behavioral: Progressive relaxation exercise — In this study, the relaxation exercises CD, which is a material created by the Turkish Psychological Association, was used. This CD consists of three parts. The first part consists of 10 minutes and this part explains the definition and purpose of deep relaxation exercise and the points to be considered during the exercise. The second part of the CD consists of 30 minutes of verbal explanation of the items of relaxation exercises accompanied by the sound of a stream. The third part consists of 30 minutes and includes only relaxation music.
  Other Names: PGE
  Arms: progressive relaxation exercises group
Other: Control group: Standart nursing care group — Routine postoperative patient care in the clinic was applied.
  Arms: Control group

SUMMARY:
This study aimed to investigate the effect of progressive relaxation exercises on the comfort and anxiety levels of patients undergoing lumbar disc herniation surgery in the neurosurgery clinic.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of progressive relaxation exercises on the comfort and anxiety levels of patients undergoing lumbar disc herniation surgery in the neurosurgery clinic.The study's data was conducted as experimental study on patients who will undergo surgery in the neurosurgery clinic of the Ministry of Health Muammer Ağım Gemlik State Hospital between March 2023 and July 2023. The sociodemographic Characteristics Questionnaire, Immobilisation Comfort Scale and State Anxiety Scale were used for data collection. The Shapiro-Wilk normality test, the t-test for the same and different groups mean and standard deviation, Pearson correlation analysis were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, elective surgery,
* Undergoing LDH surgery for the first time,
* Undergoing lumbarmicrodiscectomy surgery,
* ASA 1 and 2 classification,
* Receiving only general anaesthesia under endotracheal intubation,
* Without cognitive impairment, hearing and vision problems,
* Volunteered to participate in the study,
* Patients who did not develop any complications that would affect comfort and anxiety

Exclusion Criteria:

* 18 years of age or younger,
* With psychiatric disorders,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Comfort | Comfort levels of the patients were measured on the morning of the first postoperative day (before mobilisation)
  Measured using the "Immobilisation Comfort Scale". The total scores obtained from the scale vary between 20 and 120, and a high score indicates that the comfort is good.
Anxiety | postoperative day 1 before patients are mobilised
  Measured with "State Anxiety Scale". The state anxiety section of the state trait anxiety scale was used. In the evaluation of the scale, all items are summed and this score is subtracted from the sum of the items marked as reversed and the number 50 is added to the result. The result is the state anxiety score. The total score that can be obtained from the scale is minimum 20 and maximum 80. The increase in the score in this range indicates that the anxiety level of the individual increases.

CONTACTS AND LOCATIONS:
Overall Officials: Didem Ayhan, Associate Professor, Study Director — Bandırma Onyedi Eylül Üniversity
Locations (1):
- Gemlik Muammer Ağım State Hospital, Bursa, Gemlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No